CLINICAL TRIAL: NCT00024180
Title: A Phase I Study of Depsipeptide in Selected Hematologic Malignancies (NSC 630176)
Brief Title: FR901228 in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068898; OSU-00H0350; NCI-27
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2002-11

CONDITIONS: Leukemia; Lymphoma
Keywords: Waldenström macroglobulinemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — romidepsin

INTERVENTIONS:
Drug: romidepsin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of FR901228 in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the in vivo biologic effect of FR901228 (depsipeptide) in patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, acute myeloid leukemia, or acute lymphoblastic leukemia.
* Determine the pharmacokinetics and cellular pharmacodynamics of this drug in these patients.
* Determine any preliminary anti-tumor activity of this drug in these patients.

OUTLINE: This is a dose-decreasing, multicenter study. Patients are stratified according to disease (chronic lymphocytic leukemia and small lymphocytic lymphoma vs acute myeloid leukemia and acute lymphoblastic leukemia).

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Cohorts of 10 patients per stratum receive decreasing doses of FR901228 until the minimal active dose is determined. If 5 or more patients show clinical or biological response, the subsequent cohort is treated at a lower dose. If fewer than 5 patients respond, the subsequent cohort is treated at a higher dose.

PROJECTED ACCRUAL: A minimum of 20 patients (10 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematologic malignancies:

  * Chronic lymphocytic leukemia (CLL)
  * Small lymphocytic lymphoma (SLL) (including Waldenstrom's macroglobulinemia)
  * Acute myeloid leukemia (AML)
  * Acute lymphoblastic leukemia (ALL)
* Stratum I (CLL and SLL):

  * Received at least one prior therapy containing a purine analog OR
  * Received another form of therapy (including alkylating agents) due to history of severe autoimmune disease, requirement for chronic corticosteroid, or other contraindication to purine analog therapy
* Stratum II (AML and ALL):

  * Primary refractory or relapsed leukemia within the past year that is not amenable to curative therapy
  * OR
  * Untreated or previously treated poor-risk leukemia defined by any of the following:

    * 65 years of age and over
    * Poor-risk candidates for aggressive chemotherapy
    * Poor-risk cytogenetics (for AML, karyotype abnormalities other than t(8;21), inv(16), t(15;17))

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Stratum I only:

  * No uncontrolled autoimmune hemolytic anemia
  * No idiopathic thrombocytopenic purpura
* Stratum II only:

  * WBC no greater than 10,000/mm^3 OR
  * WBC no greater than 40,000/mm^3 that is stable for at least 1 week (may be sustained by hydroxyurea through the first week of study)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT and AST no greater than 3 times upper limit of normal

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* Ejection fraction at least 50% by MUGA
* No myocardial infarction or unstable angina within the past 6 months
* No prior unstable ventricular or supraventricular cardiac arrhythmias

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other medical or psychiatric problem that would preclude study
* Stratum I only:

  * No active infection requiring oral or IV antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 28 days since prior chemotherapy (except hydroxyurea)
* At least 6 weeks since prior nitrosoureas
* At least 8 weeks since prior UCN-01 (unless plasma UCN-01 level less than 1 uM)

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* At least 28 days since prior radiotherapy

Surgery:

* At least 28 days since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Byrd JC, Marcucci G, Parthun MR, Xiao JJ, Klisovic RB, Moran M, Lin TS, Liu S, Sklenar AR, Davis ME, Lucas DM, Fischer B, Shank R, Tejaswi SL, Binkley P, Wright J, Chan KK, Grever MR. A phase 1 and pharmacodynamic study of depsipeptide (FK228) in chronic lymphocytic leukemia and acute myeloid leukemia. Blood. 2005 Feb 1;105(3):959-67. doi: 10.1182/blood-2004-05-1693. Epub 2004 Oct 5. PMID 15466934